CLINICAL TRIAL: NCT05302661
Title: Effect of Re-education on Rebleeding Rate After Endoscopic Treatment of Esophageal and/or Gastric Varices in Patients With Liver Cirrhosis
Brief Title: Effect of Re-education on Rebleeding Rate After Endoscopic Treatment in Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20211013-Li
Record Dates: First submitted 2021-10-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Liver Cirrhosis; Esophageal Varices Bleeding; Gastric Variceal Bleeding; Bleeding
MeSH Terms: conditions — Liver Cirrhosis; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group will receive re-education after leave hospital (Experimental): The participants were randomly divided into re-education group and non re-education group according to the random number table. The re-education group will receive regular re-education not noly when they leave hospital but also after leave hospital in our preset time by telephone or wechat. The content of re-education includes diet form and diet structure,medication compliance and regularity, and recheck compliance, moderate exercise and so on
  Interventions: Behavioral: re-education
- control case group will receive no re-education after leave hospital (No Intervention): The participants were randomly divided into re-education group and non re-education group according to the random number table. without re-education group will receive regular re-education when they leave hospital.The content of re-education includes diet form and diet structure,medication compliance and regularity, and recheck compliance, moderate exercise and so on

INTERVENTIONS:
Behavioral: re-education — Contact patients by phone or wechat and guide them
  Arms: case group will receive re-education after leave hospital

SUMMARY:
A prospective, randomized controlled study on whether re-education after discharge can reduce the rebleeding rate after endoscopic treatment of esophageal and gastric varices in patients with liver cirrhosis

DETAILED DESCRIPTION:
After receiving esophageal variceal ligation and （or） gastric fundus variceal sclerotherapy, patients with outside hospitalthe rate of bleeding due to liver cirrhosis shall be re-educated outside the hospital, including diet, drugs, anticoagulation of portal vein thrombosis,regular endoscopic treatment, reexamination , nutrition, etc. The patients were divided into the first treatment group and the more thanonce treatment group according to whether they had received endoscopic treatment in the past

ELIGIBILITY:
Inclusion Criteria:

* Esophageal and / or gastric varices ；
* liver cirrhosis ；
* patients receiving endoscopic treatment (esophagogastric variceal sclerosis and/or ligation) ；
* All subjects or their guardians must sign the subject consent form before entering the test

Exclusion Criteria:

* Patients with mental illness, severe hearing loss and unable to take care of themselves ;
* ASA score ≥ grade IV at discharge ;
* Hepatic encephalopathy ≥ stage II;
* Patients with liver cancer;
* Pregnant and lactating women;
* Patients who cannot sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2022-02-19 (Actual); Primary Completion 2024-02-19 (Estimated); Study Completion 2024-02-19 (Estimated)

PRIMARY OUTCOMES:
rebleeding | 2 yeas
  rebleeding from any channel can be followed up through medical institutions or telephone

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China